CLINICAL TRIAL: NCT04506229
Title: Genetic Mechanisms Underlying SARS-CoV-2 Infection and the Impact of COVID-19 on Cognitive Function
Acronym: GenCov
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Texas Cardiac Arrhythmia Research Foundation (Other)
Responsible Party: Principal Investigator, Andrea Natale, Executive Medical Director, Texas Cardiac Arrhythmia Research Foundation
Other Study IDs: TCAI_GenCov
Record Dates: First submitted 2020-08-07; First posted 2020-08-10 (Actual); Last update posted 2020-08-27 (Actual); Status verified 2020-08

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — Exome Sequencing; Neuropsychological Tests

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COVID-19 positive
  Interventions: Genetic: Whole exome sequencing
- COVID-19 negative
  Interventions: Genetic: Whole exome sequencing

INTERVENTIONS:
Genetic: Whole exome sequencing — MoCA survey to evaluate cognitive function in COVID-19 positive cases with vs without neurological symptoms
  Other Names: Cognitive function

SUMMARY:
There is a considerable variation in the disease behavior in terms of contracting the infection, manifesting none to a range of symptoms and severity of the infection among individuals exposed to or infected with SARS-CoV-2 virus, the causative organism of COVID-19. Although the respiratory system appears to be the primary target of this virus infection, emerging evidences suggests involvement of extra-pulmonary organs including central nervous system. We aim to compare the genetic profile of individuals with vs without COVID-19 after being exposed to infected cases. Additionally, we will assess the cognitive function in covid-19 positive cases with vs. without neurological symptoms at the time of infection and 1-month follow-up using the Montreal Cognitive Assessment (MoCA) questionnaire.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female over 18 years of age at the time of enrollment
2. Have symptoms of COVID-19 (with or without hospitalization) or contact history
3. Willing to undergo nasopharyngeal swab test for viral-RNA at baseline (in non-hospitalized cases) and the MoCA survey at baseline and 1-month follow-up

Exclusion Criteria:

1. Unwilling to provide informed consent
2. MoCA score ≤17 at baseline
3. Patients with clinical diagnosis of dementia
4. Impaired consciousness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Known exposure to COVID-19 or confirmed cases of COVID-19
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2020-08-20 (Actual); Primary Completion 2021-08 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Genetic variants with vs without COVID-19 | 1 day
  Evaluate variants in the following known COVID-associated genes, ACE2R, IFITM, HLA-B 46, HLA-B 15, Toll Like Receptor and IFN-1, LIST, Perforin and mutations in Chromosome 3p21.31 along with novel genetic variants.
Cognitive function at baseline | 1 day
  Assess the cognitive status at baseline using MoCA survey in patients with vs without neurological symptoms

SECONDARY OUTCOMES:
Change in cognitive function at 1 month | 1 month
  change in the MoCA score from baseline in patients with vs without neurological symptoms
Genetic analysis | 1 day
  compare the genetic variants in patients with no or mild to moderate vs severe symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Natale, Principal Investigator — Texas Cardiac Arrhythmia Institute, St.
Locations (1):
- Texas Cardiac Arrhythmia Institute, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided